CLINICAL TRIAL: NCT05524376
Title: Regulatory Network and Diagnostic Value of Key Autophagy-related Genes in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2022-251-01
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Sepsis; Autophagy
Keywords: sepsis; autophagy
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sepsis group
  Interventions: Other: no intervention
- control group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Autophagy plays an important role in the occurrence and development of sepsis. This study aims to explore and verify the key autophagy-related genes in sepsis, then construct their regulatory networks and evaluate their potential diagnostic value, so as to provide new ideas for the diagnosis and treatment of sepsis.

DETAILED DESCRIPTION:
(1) Sepsis-related datasets GSE65682,GSE134347 and GSE134358 were downloaded from GEO database, and DEmRNA,DElncRNA and DEmiRNA were obtained by differential analysis. (2) Autophagy related genes (ARGs) were obtained from Human Autophagy Database, and ARGs in GSE65682 and GSE134347 were extracted. DEARGs were obtained by differential analysis, and GO and KEGG enrichment analysis were performed. (3) Sepsis-related genes were obtained by WGCNA analysis, and key DEARGs in sepsis were obtained by intersection with DEARGs, and then transcription factors and ceRNA regulatory network were analyzed. (4) Immune infiltration analysis was used to evaluate the distribution of immune cells in the blood of patients with sepsis, and its correlation with key DEARGs was further analyzed. (5) The diagnostic functions of key DEARGs were analyzed. (6) Peripheral blood samples from sepsis patients and healthy controls were collected and verified by RT-qPCR.

ELIGIBILITY:
Inclusion Criteria:1) over 18 years old; 2) Meeting the diagnostic criteria of Sepsis 3.0; 3) Hospital stay longer than 24 hours.

Exclusion Criteria:1) Malignant tumor; 2) Autoimmune diseases; 3) Use of immunosuppressants in the past two weeks; 4) Readmission or transfer from another ICU due to the same disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sepsis group: Eligible patients with sepsis admitted to the ICU of Sun Yat-sen Memorial Hospital of Sun Yat-sen University from September 2022 to December 2022.
  control group: Age - and sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Value of Key Autophagy-related Genes in Sepsis | October 2022
  The diagnostic functions of key DEARGs (Differential Autophagy-related Genes) were analyzed
Regulatory Network of Key Autophagy-related Genes in Sepsis | October 2022
  Key DEARGs in sepsis were analyzed for transcription factors and ceRNA regulatory network
Verified Key Autophagy-related Genes in Sepsis by RT-qPCR. | December 2022
  Peripheral blood samples from sepsis patients and healthy controls were collected and verified by RT-qPCR.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Takahashi W, Watanabe E, Fujimura L, Watanabe-Takano H, Yoshidome H, Swanson PE, Tokuhisa T, Oda S, Hatano M. Kinetics and protective role of autophagy in a mouse cecal ligation and puncture-induced sepsis. Crit Care. 2013 Jul 24;17(4):R160. doi: 10.1186/cc12839. PMID 23883625
- [Background] Aguirre A, Lopez-Alonso I, Gonzalez-Lopez A, Amado-Rodriguez L, Batalla-Solis E, Astudillo A, Blazquez-Prieto J, Fernandez AF, Galvan JA, dos Santos CC, Albaiceta GM. Defective autophagy impairs ATF3 activity and worsens lung injury during endotoxemia. J Mol Med (Berl). 2014 Jun;92(6):665-76. doi: 10.1007/s00109-014-1132-7. Epub 2014 Feb 19. PMID 24535031
- [Background] Oami T, Watanabe E, Hatano M, Sunahara S, Fujimura L, Sakamoto A, Ito C, Toshimori K, Oda S. Suppression of T Cell Autophagy Results in Decreased Viability and Function of T Cells Through Accelerated Apoptosis in a Murine Sepsis Model. Crit Care Med. 2017 Jan;45(1):e77-e85. doi: 10.1097/CCM.0000000000002016. PMID 27618275